## <u>Title</u>

Low Dose Ketamine Infusion for Comorbid Posttraumatic Stress Disorder and Chronic Pain Patients

NCT number: NCT04322968

Document Date: 10/9/2020

## STATISTICAL ANALYSIS

Statistical analyses were performed in R (R Development Core Team, 2013; version 3.5.1). Three-way repeated measures ANOVAs were conducted in order to assess differences in side effects (i.e. PRISE 20), pain symptoms (i.e. VAS, BPI-P, BPI-I), and dissociative symptoms (i.e. CADSS) by group and administered medication. Two-way repeated measures ANOVAs were conducted to assess differences in PTSD symptoms (i.e. IES-R) by medication in both the CP and CP+PTSD groups separately given predetermined differences in PTSD symptoms by group. Two-way ANOVAs were also conducted to assess the a priori primary outcomes of PTSD (IES-R) and pain (VAS) symptom change from baseline to 24 hours post infusion and the secondary outcomes of PTSD and pain symptom change from baseline to 7 days post infusion. Post-hoc analyses were conducted for all significant three-way interactions to clarify directionality of effects between and within-groups, respectively. Bonferroni corrections were used to adjust for multiple tests. Significance values for all analyses utilized a 95% confidence interval.